CLINICAL TRIAL: NCT04564170
Title: Characterization and Relationship Between Eating Disorders and Autism Spectrum Disorders.
Brief Title: Eating Disorders and Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TCA-2020-11
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Eating Disorders
Keywords: eating disorders; autism spectrum disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ED: Patients with Eating Disorders
- HC: Healthy Controls without eating disorders

SUMMARY:
This is an observational study where patients with eating disorders (ED) are compared with healthy controls without eating disorder (HC) regarding eating disorders features and autism spectrum features. Also patients will be reassessed after 5 years.

DETAILED DESCRIPTION:
The first author who suggested that eating disorders (EAD) and autism spectrum disorders (ASD) share common features was Christopher Gilberg in 1980. Currently it is known that patients with ED have social impairment, which is also a risk marker to develop ED, eating disturbances are overrepresented in ASD, ED and ASD have common behavioural features such as rigidity, perfectionism, and harm avoidance; and common cognitive profiles such as inflexibility, high attention to detail, high scores in systemizing profiles and poor results in advanced theory of mind tests. This relationship is also supported by similar neural phenotypes such as atypical structure and function in social brain regions found in both disorders.

The aim of the present study is to explore the relationship between ED and ASD traits in a sample of Spanish participants diagnosed with AN, bulimia nervosa (BN), binge-eating disorder (BED) and other eating disorders (OED). Specifically, the investigators aim to explore possible differences within the different ED and its particular transdiagnostic features in association with autistic traits.

The sample will consist of 90 patients with ED and 45 healthy controls (HC) without any current or lifetime history of mental disorder, both groups will be compared regarding ED and ASD features. Also patients will be reassessed in a 5 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Being Diagnosed with ED

Exclusion Criteria:

* language or intellectual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ED and HC without ED.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Autism Spectrum Quotient | one year
  A self report measure of autism traits. Its values range from 0 to 50. Higher scores mean higher autistic traits.
Eating Disorders Inventory | one year
  A self report measure of Eating Disorders characteristics. Its values range from 0 to 192, higher values mean higher eating disorders symptomatology.

SECONDARY OUTCOMES:
Bulimic Investigatory Test Edinburgh | one year
  A self report measure of bulimic symptoms where higher scores mean more bulimic symptomatology. Scores range from 0 and 78.
Quality of Life Enjoyment and Satisfaction Questionnaire | one year
  The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. Its values range from 93 to 465. Higher values mean higher quality of life.
Beck Depression Inventory | one year
  a self report measure of depression symptomatology. Scores rang form 0 to 63, higher scores mean more depressive symptomatology.
Scale Unawareness of Mental Disorders. | one year
  A scale to asess awareness of mental disorders where higher punctuation mean higher levels of unawareness of the disorder. Scores range from 20 to 100.
Body Shape Questionnaire | one year
  A a self-report measure of the body shape preoccupations typical of bulimia nervosa and anorexia nervosa. Higher scores mean higher concern with shape. Score range from 34 to 204.
Rosenberg Self -Esteem Scale | one year
  A self report measure of self esteem. Its scores range from 10 to 40 where higher scores mean higher self -esteem
State Trait Anxiety Inventory | one year
  A self report measure of anxiety symptomatology. It has two scores one for state of anxiety and another for trait of anxiety, each subscale values range from 0 to 60, higher scores mean higher state or trait of anxiety.
Inventory of interpersonal problems personality disorder | one year
  A self report measure which is used to identify problems associated with particular personality disorders. Its values range from 0 to 256, higher scores mean higher interpersonal problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Carmona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atienza, F., Moreno, Y., & Balaguer, I. (2000). Escala de autoestima de Rosenberg. Recuperado de: https://www. uv. es/uipd/cuestionarios/accesolibre/EAR.
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). BDI-II: Beck depression inventory. Pearson.
- [Background] Bentz M, Jepsen JRM, Pedersen T, Bulik CM, Pedersen L, Pagsberg AK, Plessen KJ. Impairment of Social Function in Young Females With Recent-Onset Anorexia Nervosa and Recovered Individuals. J Adolesc Health. 2017 Jan;60(1):23-32. doi: 10.1016/j.jadohealth.2016.08.011. Epub 2016 Oct 27. PMID 28341015
- [Background] Cooper, P. J., Taylor, M. J., Cooper, Z., & Fairbum, C. G. (1987). The development and validation of the Body Shape Questionnaire. International Journal of eating disorders, 6(4), 485-494.
- [Background] First, M. B. (2015). DSM-5 : Manual de diagnóstico diferencial (DSM-V). Editorial Médica Panamericana.
- [Background] Huke V, Turk J, Saeidi S, Kent A, Morgan JF. Autism spectrum disorders in eating disorder populations: a systematic review. Eur Eat Disord Rev. 2013 Sep;21(5):345-51. doi: 10.1002/erv.2244. Epub 2013 Jul 31. PMID 23900859
- [Background] Khalsa SS, Portnoff LC, McCurdy-McKinnon D, Feusner JD. What happens after treatment? A systematic review of relapse, remission, and recovery in anorexia nervosa. J Eat Disord. 2017 Jun 14;5:20. doi: 10.1186/s40337-017-0145-3. eCollection 2017. PMID 28630708
- [Background] Nielsen S, Anckarsater H, Gillberg C, Gillberg C, Rastam M, Wentz E. Effects of autism spectrum disorders on outcome in teenage-onset anorexia nervosa evaluated by the Morgan-Russell outcome assessment schedule: a controlled community-based study. Mol Autism. 2015 Mar 8;6:14. doi: 10.1186/s13229-015-0013-4. eCollection 2015. PMID 25774282
- [Background] Oldershaw A, Treasure J, Hambrook D, Tchanturia K, Schmidt U. Is anorexia nervosa a version of autism spectrum disorders? Eur Eat Disord Rev. 2011 Nov-Dec;19(6):462-74. doi: 10.1002/erv.1069. Epub 2011 Jan 30. PMID 21280165
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R. E., Vagg, P. R., & Jacobs, G. A. (1970). Manual for the state-trait inventory. Consulting Psychologists, Palo Alto, California.
- [Background] Westwood H, Eisler I, Mandy W, Leppanen J, Treasure J, Tchanturia K. Using the Autism-Spectrum Quotient to Measure Autistic Traits in Anorexia Nervosa: A Systematic Review and Meta-Analysis. J Autism Dev Disord. 2016 Mar;46(3):964-77. doi: 10.1007/s10803-015-2641-0. PMID 26542816